CLINICAL TRIAL: NCT04025307
Title: A Multi-centre, Open-label, Phase I Trial of bacTRL-IL-12 in Adult Subjects With Advanced, Treatment-refractory Solid Tumours
Brief Title: Phase I Trial of bacTRL-IL-12 in Adult Subjects With Advanced, Treatment-refractory Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bacTRL-IL-12-001
Record Dates: First submitted 2019-07-11; First posted 2019-07-18 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Cancer - Solid Tumours

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bacTRL-IL-12 (Experimental): single-dose, 1 mL IV infusion of bacTRL-IL-12
  Interventions: Drug: bacTRL-IL-12

INTERVENTIONS:
Drug: bacTRL-IL-12 — bacTRL-IL-12 is a live, genetically modified Bifidobacterium longum (B longum), for administration via IV infusion. The probiotic bacteria selectively colonize solid tumour tissues and are engineered to deliver genetic material encoding the pro-inflammatory transgene Interleukin-12 (IL-12). Plasmid DNA encoding the IL-12 transgene is delivered to the patient's cells within the tumor microenvironment, whereupon IL-12 is expressed to stimulate local and systemic anti-tumour immune responses.

SUMMARY:
This study is as an open-label study to be conducted at multiple study centres across New Zealand and Australia designed to characterise the safety, tolerability and preliminary assessment of the anti-tumour efficacy of bacTRL-IL-12 after intravenous (IV) infusion.

The study will consist of a screening period (Day -14 to Day -2), treatment and observation (Day 1 to Day 22), safety follow-up period (Day 28 to Day 31), and efficacy follow-up period (until progression, death, revocation of consent, or lost to follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years or older);
2. Capable of providing informed consent;
3. Advanced and/or metastatic, histologically-documented, measurable (per iRECIST) solid tumours for which there are no other standard therapy options available that are acceptable to the subject;
4. Eastern Cooperative Oncology Group status of 0 or 1;
5. Adequate haematological status (regardless of transfusions) defined as:

   * Absolute neutrophil count ≥ 1.5 x 109/L;
   * Platelets ≥ 100 x 109/L;
   * Haemoglobin ≥ 9g/dL;
6. Adequate renal function, defined as estimated serum creatinine clearance > 45mL/minute calculated using Cockcroft-Gault equation
7. Adequate coagulation function, defined as:

   * International Normalised Ration <1.5 x upper limit of normal (ULN) for that laboratory
   * Partial thromboplastin time <1.5 x ULN
   * Exception: monitoring parameters must be within therapeutic range for subjects receiving anti-coagulation therapy
8. Adequate hepatic function, defined as:

   * Total bilirubin < 1.5 x ULN unless considered due to Gilbert's disease;
   * Alanine aminotransferase and aspartate aminotransferase < 1.5 x ULN or < 3 x ULN with documented liver metastases;
9. Recovery from the toxicities of previous anti-cancer drugs or radiotherapy to Grade 0 or 1 (or to baseline if condition was pre-existing);
10. A female subject is eligible to participate if she in not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

    * Not of childbearing potential, defined as surgically sterile (documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or postmenopausal *no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is sufficient);
    * Of childbearing potential and agrees to use a highly effective method of contraception consistently during the treatment period and for at least 60 days after that dose of study treatment;
11. A male subject with a female partner of childbearing potential is eligible to participate if he agrees to use acceptable contraception during the treatment period and for at least 60 days after the last dose of study treatment and refrains from donating sperm during this period;
12. Agree to increase oral sugar intake during the treatment period.

Exclusion Criteria:

1. Presence or history of brain metastases or abscess;
2. Presence of known or suspected ongoing ischemia of non-tumor tissues that may be inadvertently colonized by bacteria including:

   * Ischemic peripheral vascular disease, myocardial infarction within the past 6 months;
   * Congestive heart failure > class II New York Heart Association;
   * Unstable angina (anginal symptoms at rest) or new onset angina (commenced within the last 3 months);
   * Patent foramen ovale;
   * Prior history or current bacterial endocarditis,
   * Existing thrombus (either arterial or venous) as well as known history of deep vein thrombosis, permanent pacemakers, automated implantable cardioverter-defibrillators, left ventricular assist devices, or other intravascular cardiac device, known arteriovenous malformations;
   * Cerebrovascular event, including transient ischemic attacks within the past 6 months;
3. An artificial implant that cannot be easily removed (e.g., heart valves, prosthetic hips or knees, or other devices) that could allow inadvertent bacterial colonization;
4. Abnormal fluid collections (e.g. ascites and/or pericardial and/or pleural effusions) that could allow inadvertent bacterial colonization;
5. Has tumor masses immediately adjacent to, and/or with infiltration into, large arteries, veins or vessels;
6. Bacteremia and/or abscess and/or treatment with systemic (oral or IV) antibiotics within 4 weeks prior to dosing;
7. Anticipated exposure to systemic antibiotics within 4 weeks of dosing;
8. Positive for human immunodeficiency virus, hepatitis B or hepatitis C at screening;
9. Treatment with radiation therapy to a visceral organ or tumors within 2 weeks prior to dosing;
10. Treatment with any programmed cell death protein-1 and/or programmed cell death ligand 1 inhibiting agent within 2 weeks prior to dosing;
11. Treatment with any investigational agent for treatment of cancer or related comorbidity within 4 weeks prior to dosing;
12. Treatment with any chemotherapy or major surgery within 6 weeks prior to dosing;
13. History of allergic reactions attributed to compounds of similar chemical or biologic composition to agent(s) or other agents used in study;
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune disorder, or psychiatric illness/social situations that would limit compliance with study requirements;
15. Any other reason that, in the opinion of the investigator and/or sponsor, precludes the subject from participating in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events according to NCI CTCAE | day 31 safety follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Monash Medical Centre, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No